CLINICAL TRIAL: NCT00791674
Title: Sleep Disordered Breathing in Patients With Chronic Pain and Long Term Opiate Therapy
Brief Title: Opiate Sleep Disordered Breathing Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Adelaide Institute for Sleep Health (Other)
Collaborators: Flinders Medical Centre (Other Government)
Responsible Party: Dr.Anand Rose, Adelaide Institute of Sleep Health
Other Study IDs: 50/07
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2008-11-14 (Estimated); Status verified 2008-11

CONDITIONS: Sleep Apnea
Keywords: Opiates; sleep apnea; ventilatory failure
MeSH Terms: conditions — Sleep Apnea Syndromes; Hypoventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Lay title: A study of breathing pauses during sleep in patients on long term opiates.

Sleep apnoea is a term which refers to frequent breathing pauses during sleep. Breathing can stop at night due to the upper airway collapsing (Obstructive sleep apnoea)or reduced signals from the brain driving breathing (central sleep apnoea). Clinical observation has noticed that patients on opiates have an increase in sleep apnoea.

Hypothesis: This study looks at the relationship of opiates (when used for patients chronic pain) and the occurrence of sleep apnoea. It is expected that there will be an increase in sleep apnoea (particularly of the central variant) particularly in patients on long term opiates.

DETAILED DESCRIPTION:
The purpose for this study is to test the hypothesis that sleep disordered breathing is more prevalent amongst a group of patients on high dose opiates for chronic pain.

Aims

1. To define the prevalence of sleep disordered breathing in a group of patients on oral morphine for chronic pain.
2. To determine the prevalence of respiratory failure in this cohort of patients. Patients on long term opiates (>6 months) from an outpatient pain clinic population on long acting morphine formulations > 40 mg/day, Oxycontin 30 mg/day, and Methadone > 20 mg/day were prospectively recruited. Home polysomnograms were done on them. During their clinical review they have spirometry, arterial blood gases, psychomotor vigilance tests done on them.

ELIGIBILITY:
Inclusion Criteria:

* Patients on long acting Morphine >40mg/day, Oxycontin >30mg/day, and Methadone >20mg/day were contacted.
* Stable opiate dose for 2 weeks
* Lives within 80KM of FMC

Exclusion Criteria:

* Significant CCF/CVA
* Severe COPD
* Major Psychiatric illness
* History of substance abuse in the last 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pain clinic outpatients were contacted if they were on the specified doses (
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2007-12

PRIMARY OUTCOMES:
Prevalence of sleep disordered breathing in patients on long term opiates. | 18 months

SECONDARY OUTCOMES:
Prevalence of ventilatory failure in this cohort | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Anand R Rose, MD,FRACP, Principal Investigator — Adelaide Institute of Sleep Health; Doug McEvoy, MD, FRACP, Study Director — Adelaide Institute of Sleep Health, Repatriation General Hospital
Locations (2):
- Australia (2):
  - Pain Management Unit, Flinders Medical Centre, Bedford Park, South Australia
  - Adelaide Institute of Sleep Health, Repatriation General Hospital,, Daw Park, South Australia